CLINICAL TRIAL: NCT04990232
Title: Personalized Immunotherapy in Sepsis: a Multicentre and Multinational, Double-blind, Double-dummy Randomized Clinical Trial
Brief Title: Personalized Immunotherapy in Sepsis
Acronym: ImmunoSep
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ImmunoSep
Record Dates: First submitted 2021-07-29; First posted 2021-08-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: multicentre and multinational, double-blind, double-dummy randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Placebo Comparator): Patients will receive the standard type of treatment decided by the attending physicians. They will also receive 20ml (10ml for patients with creatinine clearance lower than 30ml/min) intravenous (IV) 0.9% saline (N/S) three times daily (every eight hours) for 15 days and 0.5 ml subcutaneous (sc) 1ml 0.9% N/S every other day for a total of 15 days.
  Interventions: Drug: Placebo
- Immunotherapy (Experimental): Patients will receive the standard type of treatment decided by the attending physicians. They will also receive IV anakinra 200 mg three times daily (every eight hours) or sc rhIFNγ 100 μg once every other day. More precisely, patients randomized for hyper-inflammation will receive anakinra three times daily (every eight hours) for 15 days and sc 0.5 ml N/S 0.9% every other day for 15 days. Patients having immunoparalysis will receive IV 20 ml N/S 0.9% (10ml for patients with creatinine clearance lower than 30ml/min) three times daily (every eight hours) for 15 days and sc rhIFNγ every other day for 15 days. Especially for patients with creatinine clearance lower than 30 ml/min anakinra will be given half dose (i.e. 100 mg three times daily). Creatinine clearance is calculated by the Cockcroft Gault equation [(140-age in years)/ (72 x serum creatinine in mg/dl) for men; this is multiplied by 0.85 for women.
  Interventions: Drug: Anakinra or rhIFNγ

INTERVENTIONS:
Drug: Anakinra or rhIFNγ — In hyper-inflammation anakinra three times daily (every eight hours) for 15 days and sc 0.5 ml N/S 0.9% every other day for 15 days. In immunoparalysis IV 20 ml N/S 0.9% (10ml for patients with creatinine clearance lower than 30ml/min) three times daily (every eight hours) for 15 days and sc rhIFNγ every other day for 15 days.
  Other Names: Imukin; Kineret
  Arms: Immunotherapy
Drug: Placebo — 20ml (10ml for patients with creatinine clearance lower than 30ml/min) intravenous (IV) 0.9% saline (N/S) three times daily (every eight hours) for 15 days and 0.5 ml subcutaneous (sc) 1ml 0.9% N/S every other day for a total of 15 days
  Arms: Standard of care

SUMMARY:
Αim of ImmunoSep is to assess whether personalized adjunctive immunotherapy directed against a state of either fulminant hyper-inflammation or immunoparalysis is able to change sepsis outcomes. Patients will be selected by a panel of biomarkers and laboratory findings and will be allocated to placebo or immunotherapy treatment according to their needs.

DETAILED DESCRIPTION:
Sepsis is a life-threatening organ dysfunction that results from the dysregulated host response to an infection. Accumulating knowledge suggests that there is a spectrum of dysregulation in this response. On the one end of this spectrum there are patients whose immune response is characterized by fulminant hyper-inflammation. On the other end of this spectrum there are patients whose immune response is characterized by immunoparalysis. The majority of patients are situated between these two extremes. The primary hypothesis of the ImmunoSep trial is to recognize both ends of this spectrum and to administer adjunctive therapy aiming to modulate the sepsis-associated hyper-inflammation or immunoparalysis. It is anticipated that with this strategy patients' organ dysfunctions be improved.

During the last years the Hellenic Sepsis Study Group (HSSG) managed to develop ferritin as the diagnostic tool for the recognition of patients with fulminant sepsis-associated hyper-inflammation. This was done by analysis of 5,121 patients split into a test and a validation cohort and by also studying a confirmation cohort coming from Sweden. Patients were classified according to the criteria for the macrophage activation syndrome developed by the American College of Rheumatology; approximately 4% of patients with sepsis have fulminant hyper-inflammation or macrophage activation-like syndrome (MALS) that is an independent clinical condition associated with short-term 10-day mortality. Serum ferritin greater than 4,420 ng/ml had sensitivity 97.1% and negative predictive value 98% for the diagnosis. More than 25 years ago one randomized clinical trial (RCT) was conducted where patients with severe sepsis were randomly assigned to blind treatment with placebo or with the recombinant human interleukin-1 receptor antagonist anakinra. The trial failed to disclose any benefit of anakinra on 28-day mortality. However, a recent post-hoc analysis revealed that patients who had signs of macrophage activation syndrome had significant 30% survival benefit by anakinra treatment.

The immunoparalysis of sepsis is associated with at least 50% risk of death in the subsequent 28 days. There is evidence from preclinical studies and from the endotoxin challenge model in human volunteers that this can be reversed using recombinant human interferon gamma (rhIFNγ). rhIFNγ was administered in nine patients with septic shock in a small open-label clinical trial without placebo comparator; reversal of immunoparalysis was achieved.

It is important to recognize patients with sepsis complicated either with MALS or with immunoparalysis and administer anakinra or rhIFNγ respectively as a potentially beneficial intervention. To this end, a smaller-scale trial was conducted in Greece that was aiming to the personalized management of septic shock. The acronym of this trial was PROVIDE. PROVIDE was conducted between December 2017 and December 2019 in 14 study sites in Greece under the auspices of the European Shock Society. In the PROVIDE trial patients with septic shock due to lower respiratory tract infection, acute cholangitis, or primary bacteremia, were screened on two consecutive days for laboratory signs of fulminant hyper-inflammation or immunoparalysis. Results showed that one single measurement of serum ferritin and the number of human leukocyte antigen-DR (HLA-DR) on monocytes can efficiently classify patients. More precisely, ferritin 4,420 ng/ml diagnoses MALS; and a combination of ferritin >4,420 ng/ml and HLA-DR less than 5000 molecules/monocyte diagnose imunoparalysis. Patients were randomized into double-dummy blind treatment with placebo if randomly assigned to the standard-of-care arm and with anakinra/recombinant human interferon-gamma (rhIFNγ) if randomly assigned to the immunotherapy arm. Thirty-six patients were enrolled and preliminary results derived from the PROVIDE trial further corroborate the use of anakira/rhIFNγ as an innovative, personalized adjunct therapy for sepsis but one larger-scale study with larger number of patients is needed in order to validate findings.

ImmunoSep is a randomized placebo-controlled phase 2 clinical trial with a double-dummy design where the effect of personalized immunotherapy in patients with sepsis and either fulminant hyper-inflammation or immunoparalysis is studied. Hyper-inflammation is considered as a more direct life-threatening manifestation of sepsis than immunoparalysis; for that reason patients with lab findings of both immune states are allocated to the hyper-inflammation treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years.
* Both genders.
* In case of women, unwillingness to become pregnant during the study period.
* Written informed consent provided by the patient or by one first-degree relative/spouse in case of patients unable to consent.
* Community-acquired pneumonia (CAP) or hospital-acquired pneumonia (HAP) or ventilator-associated pneumonia (VAP) or primary bacteremia (BSI).
* Sepsis defined by the Sepsis-3 definitions. More precisely, sepsis is defined as the presence of total SOFA (sequential organ failure assessment score) equal to 2 or more for patients who are admitted with infection at the emergency department OR as any increase of admission SOFA by 2 or more points for patients already hospitalized.
* Patients with signs of fulminant hyper-inflammation or sepsis-associated immunoparalysis as defined by ferritin and Quantibrite. Since the state of hyper-inflammation is considered more life-threatening than the state of immunoparalysis, patients with lab findings of both immune states are allocated to treatment targeting hyper-inflammation. It is explicitly stated that patients diagnosed with novel Coronavirus-2 infection (COVID-19) may participate only in the fulminant hyper-inflammation arm
* Time from classification into sepsis by the Sepsis-3 definitions and start of blind intervention less than 72 hours.

Exclusion Criteria:

* Age below 18 years.
* Denial for written informed consent.
* Acute pyelonephritis or intraabdominal infection, meningitis or skin infection.
* Any stage IV malignancy.
* Neutropenia defined as an absolute neutrophil count lower than 1,500/mm3.
* Any 'do not resuscitate' decision in the hospital.
* In the case of BSI, patients with blood cultures growing coagulase-negative staphylococci or skin commensals or catheter-related infections cannot be enrolled.
* Active tuberculosis (TB) as defined by the co-administration of drugs for the treatment of TB.
* Infection by the human immunodeficiency virus (HIV).
* Any primary immunodeficiency.
* Oral or intravenous intake of corticosteroids at a daily dose equal or greater than 0.4 mg/kg prednisone or greater the last 15 days.
* Any anti-cytokine biological treatment the last one month.
* Medical history of systemic lupus erythematosus.
* Medical history of multiple sclerosis or any other demyelinating disorder.
* Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-04-27 (Actual)

PRIMARY OUTCOMES:
Mean total Sequential Organ Failure Assessment score | 9 days
  Difference in the mean total Sequential Organ Failure Assessment score between the two arms

SECONDARY OUTCOMES:
28-day mortality | 28 days
  Difference in mortality between the two arms
90-day mortality | 90 days
  Difference in mortality between the two arms
Mean total Sequential Organ Failure Assessment score | 15 days
  Difference in the mean total Sequential Organ Failure Assessment score between the two arms
Reversal of hyper-inflammation (decrease of ferritin) or immunoparalysis (increase of Quantibrite) | 15 days
  Difference in percentage of patients between the two arms with any at least 15% decrease of the baseline serum ferritin (if in hyper-inflammation) and with any Quantibrite to above 8,000 AB/C with serum ferritin below 4,420 ng/ml (if in sepsis-associated immunoparalysis)

OTHER OUTCOMES:
Resolution of infection-reversal of all signs and symptoms of the initial infection | 15 days
  Difference in percentage of patients with resolution of the initial infection between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Evagelos Giamarellos-Bourboulis, MD, PhD, Study Chair — Hellenic Institute for the Study of Sepsis
Locations (35):
- Intensive Care Unit, Jena University Hospital, Jena, Jena, Germany
- Greece (29):
  - Intensive Care Unit, Alexandroupolis University Hospital, Alexandroupoli, Alexandroupolis
  - 1st Department of Pulmonary Medicine and Intensive Care Unit, Athens, Athens
  - 3rd University Department of Internal Medicine, General Hospital of Chest Diseases of Athens SOTIRIA, Athens, Athens
  - New Intensive Care Unit, SOTIRIA Athens General Hospital of Chest Diseases, Athens, Athens
  - 2nd Department of Critical Care Medicine, ATTIKON University Hospital, Athens, Haidari
  - Intensive Care Unit, Ioannina University Hospital, Ioannina, Ioannina
  - Intensive Care Unit, Center for Accident Rehabilitation (KAT) of Athens, Athens, Kifissia
  - Department of Internal Medicine, Larissa University Hospital, Larissa, Larissa
  - Intensive Care Unit, TZANEIO Piraeus General Hospital, Piraeus, Piraeus
  - Intensive Care Unit, 424 General Military Training Hospital, Thessaloniki, Thessaloniki
  - 1ST Department of Internal Medicine, Evangelismos General Hospital, Athens
  - General Hospital of Athens LAIKO - Intensive Care Unit, Athens
  - Intensive Care Unit of Center for Respiratory Failure, General Hospital of Chest Diseases of Athens SOTIRIA, Athens
  - 4th Department of Internal Medicine, "Attikon" University Hospital, National and Kapodistrian University of Athens, Medical School, Athens
  - Intensive Care Unit, General Hospital ASKLEPIEIO Voulas, Athens
  - 2nd Department of Internal Medicine, Attikon University Hospital, Athens
  - 5th Department of Internal Medicine, Evangelismos General Hospital, Athens
  - General Oncological Hospital of Kifisia Oi Agioi Anargyroi - Clinic of Intensive Care and Pulmonary Diseases Department of Nursing, University of Athens, Athens
  - Greece Intensive Care Unit General Hospital of Athens Korgialeneio, Athens
  - Intensive Care Unit, "Latsio", Thriasio Elefsis General Hospital, Elefsina
  - Greece Intensive Care Unit University General Hospital of Heraklion, Heraklion
  - General Hospital of Karditsa Intensive Care Unit, Karditsa
  - Intensive Care Unit, "Koutlimbaneio & Triantafylleio" Larissa General Hospital, Larissa
  - Intensive Care Unit, Agios Dimitrios General Hospital, Thessaloniki
  - Intensive Care Unit, G. Gennimatas General Hospital, Thessaloniki
  - Intensive Care Unit, Theageneio Oncological Hospital of Thessaloniki, Thessaloniki
  - Intensive Care Unit, Ippokrateion General Hospital, Thessaloniki
  - Department of Anesthesiology and Intensive Care Medicine, University General Hospital of Thessaloniki AHEPA, Thessaloniki
  - General Hospital of Thessaloniki, Papageorgiou- Intensive Care Unit, Thessaloniki
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Rome, Italy
- Netherlands (2):
  - Department of Internal Medicine and Infectious Diseases, Amsterdam Medical Center, Amsterdam, Amsterdam
  - Intensive Care Unit, University Medical Center Radboud, Nijmegen, Nijmegen
- Infectious Diseases Department, "Iuliu Hatieganu'' University of Medicine and Pharmacy Cluj-Napoca, Cluj-Napoca, Cluj-Napoca, Romania
- Intensive Care Unit, Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All data will be available within published manuscript. Deidentified patient data can be requested to Sponsor and shared after approval for purposed approved by Sponsor.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon publication of manuscript related to this study
Access Criteria: After contact with sponsor (egiamarel@med.uoa.gr)

REFERENCES:
- [Derived] Giamarellos-Bourboulis EJ, Kotsaki A, Kotsamidi I, Efthymiou A, Koutsoukou V, Ehler J, Paridou A, Frantzeskaki F, Muller MCA, Pickkers P, Meylan S, Nikolopoulos I, Lupse M, Gavala A, Vlachogianni G, Solomonidi N, Alevizou A, Kondili E, Antoniadou E, Nakou M, Markou N, Hatziagelaki E, Prekates A, Komnos A, Bakkerus L, Slim MA, Dalekos GN, Karapanagiotou A, Ktena S, De Pascale G, Koulouras V, Psarrakis C, Massa E, Dakou K, Pazvanti C, Ioakeimidou A, Tsangaris I, Antonakos N, Vlaar APJ, Anisoglou S, Calandra T, Papaioannou V, Myrianthefs P, Patrani M, Alamanos I, Antonelli M, van der Meer JWM, van der Poll T, Wiersinga WJ, Ntaganou M, Gkeka E, Bauer M, Mouloudi E, Netea MG; ImmunoSep Study Group. Precision Immunotherapy to Improve Sepsis Outcomes: The ImmunoSep Randomized Clinical Trial. JAMA. 2025 Dec 8:e2524175. doi: 10.1001/jama.2025.24175. Online ahead of print. PMID 41359996
- [Derived] Giamarellos-Bourboulis EJ, Dimopoulos G, Flohe S, Kotsaki A, van der Poll T, Skirecki T, Torres A, Netea MG. THE EUROPEAN SHOCK SOCIETY MEETS THE IMMUNOSEP CONSORTIUM FOR PERSONALIZED SEPSIS TREATMENT. Shock. 2023 Mar 1;59(3S Suppl 1):21-25. doi: 10.1097/SHK.0000000000001955. Epub 2022 Jul 24. PMID 36867758
- [Derived] Kotsaki A, Pickkers P, Bauer M, Calandra T, Lupse M, Wiersinga WJ, Meylan S, Bloos F, van der Poll T, Slim MA, van Mourik N, Muller MCA, van Vught L, Vlaar APJ, de Nooijer A, Bakkerus L, Weis S, Antonakos N, Netea MG, Giamarellos-Bourboulis EJ. ImmunoSep (Personalised Immunotherapy in Sepsis) international double-blind, double-dummy, placebo-controlled randomised clinical trial: study protocol. BMJ Open. 2022 Dec 20;12(12):e067251. doi: 10.1136/bmjopen-2022-067251. PMID 36600424